CLINICAL TRIAL: NCT06256653
Title: A Randomised, Double-blinded, Placebo- Controlled, Parallel Study, to Assess the Effect of a Whole Fruit Powder on Gut Microbiome Function on Overweight & Obese Adults
Brief Title: Assess the Effect of a Whole Fruit Powder on Gut Microbiome Function on Overweight & Obese Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Collaborators: U.S. Highbush Blueberry Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AFCRO-175
Record Dates: First submitted 2024-01-16; First posted 2024-02-13 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-03

CONDITIONS: Obesity; Overweight and Obesity
Keywords: Gut Microbiome; Obesity; Overweight; Gut Permeability
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Intervention Model Description: Randomised, double-blinded, placebo-controlled, parallel study in overweight and obese adults.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blinding of both study team and Participants will be ensured by only providing access to the randomisation list to the science and quality team which is stored in the quality drive. The relationship between the randomisation number and the group assignment will be unknown to the Participants, clinical study team, and the Sponsor, i.e., the study will be double-blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Freeze-dried Blueberries (Experimental): Participants will be provided with an 8-week supply of study product (freeze-dried blueberry) to be consumed daily.
  Interventions: Dietary Supplement: Freeze-dried blueberries
- Maltodextrin, Glucose, Fructose and Sucrose Placebo (Placebo Comparator): Participants will be provided with an 8-week supply of placebo product (maltodextrin, glucose 31%, fructose 30%, sucrose 0%; produced as a purple powder, with blueberry aromatics generated from natural (non-anthocyanin) and artificial colour and flavourings) to be consumed daily.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Freeze-dried blueberries — * Participants will be supplied with an 8-week supply of Study Product and instructions of dosing.
  * Participants will be instructed to mix one sachet of the Study Product either to breakfast, or dessert, or mixed with yoghurt daily for the next 56 days, starting on the same day, Day 1.
  * Additional product will be supplied in case of delay of study visit or loss of Study Product.
  * Participants will be provided with a stool collection kit and instructions for collecting and storing. Participants will collect stool samples at home, within 48 hours prior to their visit but preferably the morning, of their scheduled visit and bring it to the clinic.
  * Participants will be provided with a urine collection kit and instructions for collecting and storing.
  Arms: Freeze-dried Blueberries
Dietary Supplement: Placebo — * Participants will be supplied with an 8-week supply of Placebo Product and instructions of dosing.
  * Participants will be instructed to mix one sachet of the Placebo Product either to breakfast, or dessert, or mixed with yoghurt daily for the next 56 days, starting on the same day, Day 1.
  * Additional product will be supplied in case of delay of study visit or loss of Placebo Product.
  * Participants will be provided with a stool collection kit and instructions for collecting and storing. Participants will collect stool samples at home, within 48 hours prior to their visit but preferably the morning, of their scheduled visit and bring it to the clinic.
  * Participants will be provided with a urine collection kit and instructions for collecting and storing.
  Arms: Maltodextrin, Glucose, Fructose and Sucrose Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the effect of freeze-dried blueberry powder on the gut microbiome in overweight and obese adults. The main question[s] it aims to answer are:

* Does the supplementation of freeze-dried blueberry powder reduce the risk of obesity or lower the weight of people with a high BMI?
* Does freeze-dried blueberry powder alter the gut microbiome function? Participants will;
* Mix one sachet of Study Product (freeze-dried blueberry powder/placebo) into breakfast/dessert/yoghurt daily for 56 days during the intervention phase.
* Partake in 4 site visits over the 14-week period, including an initial screening visit and a follow-up visit after the intervention phase.

Researchers will compare the effect of freeze-dried blueberry powder with a placebo in a population comprising overweight and obese adults to see if the gut microbiome is altered and if there is a change in body composition.

DETAILED DESCRIPTION:
Definition: Extended description of the protocol, including more technical information (as compared to the Brief Summary), if desired. Do not include the entire protocol; do not duplicate information recorded in other data elements, such as Eligibility Criteria or outcome measures. For Patient Registries: Also describe the applicable registry procedures and other quality factors (for example, third party certification, on-site audit). In particular, summarize any procedures implemented as part of the patient registry, including, but not limited to the following:

* Quality assurance plan that addresses data validation and registry procedures, including any plans for site monitoring and auditing.
* Data checks to compare data entered into the registry against predefined rules for range or consistency with other data fields in the registry.
* Source data verification to assess the accuracy, completeness, or representativeness of registry data by comparing the data to external data sources (for example, medical records, paper or electronic case report forms, or interactive voice response systems).
* Data dictionary that contains detailed descriptions of each variable used by the registry, including the source of the variable, coding information if used (for example, World Health Organization Drug Dictionary, MedDRA), and normal ranges if relevant.
* Standard Operating Procedures to address registry operations and analysis activities, such as patient recruitment, data collection, data management, data analysis, reporting for adverse events, and change management.
* Sample size assessment to specify the number of participants or participant years necessary to demonstrate an effect.
* Plan for missing data to address situations where variables are reported as missing, unavailable, non-reported, uninterpretable, or considered missing because of data inconsistency or out-of-range results.
* Statistical analysis plan describing the analytical principles and statistical techniques to be employed in order to address the primary and secondary objectives, as specified in the study protocol or plan.

Randomised, double-blinded, placebo-controlled, parallel study in overweight and obese adults.

* Screening phase: 14 days
* Intervention phase: 56 days
* Follow-up phase: 28 days

Participants will be provided with an 8-week supply of product (60 sachets) at Visit 2 and instructed to consume one sachet per day for eight-weeks. Participants will be recruited via an initial pre-screening questionnaire.

Visit 1 - Screening

* Participants will receive oral and written information about the study and be allowed to ask questions, sign the informed consent document, Inclusion and exclusion criteria will be reviewed, Demographic, health, and lifestyle data will be collected.
* Participants will be provided with a stool collection kit and a urine collection kit and instructions for collecting and storing.

Visit 2 - Day 1

- Participant's continued consent to study procedures will be confirmed. Inclusion/exclusion criteria will be reviewed. Concomitant medication/supplements will be recorded. Full anthropometrics taken. Participants will return their collected stool samples and samples will be stored for further analysis. Fasting blood samples will be collected for safety analysis and for blood markers/metabolites.

Participants will be randomised into one of the two treatment groups as follows, but will be blinded as to which group they are in:

* Group 1: Freeze-dried blueberry powder
* Group 2: Placebo
* Participants will be supplied with an 8-week supply of Study Product and instructions of dosing.

Participants will be provided with a stool collection kit and a urine collection kit and instructions for collecting and storing.

Visit 3 - Day 57

Participants will return to the study site at day 57, having completed the intervention phase of the study. Participants will have fasted overnight for at least 10-hours. The following procedures will be carried out: Participant's continued consent to study procedures will be confirmed. Anthropometrics taken. Adverse events will be recorded. Participants will return their collected stool sample and sample will be stored for further analysis. Fasting blood samples will be collected for safety analysis and for blood markers/metabolites. Participants will return any unused Study Product and compliance will be assessed. Participants will collect 5-hour urine sample on-site.

Visit 4 - Day 84 (Follow-up Phase)

- Concomitant medication/supplements will be recorded. Anthropometrics taken. Adverse events will be recorded. Participants will return their collected stool samples and will be stored for

further analysis. A fasting blood sample will be collected. Participants will return with the 24 h urine collected at home the day prior of their visit.

Participants have the right to withdraw from the study at any time for any reason, without giving a reason and without penalty or loss of benefits they are entitled to.

Data processing & Management

Data required for the analysis will be acquired and transferred electronically to a central database by means of an Electronic Data Capture system (the "EDC-tool"). The EDC-tool will comprise an eCRF, designed specifically for the present study. High security standards for the transfer and storage of study data are guaranteed using technologies such as encrypted data transfer, firewalls, and periodic backup to protect centrally stored data. The eCRF is based on the electronic data capture system developed by Clindox, which is fully compliant with and a Gold Member of the Clinical Data Interchange Standards Consortium. The eCRF will be hosted on a dedicated validated stand-alone server placed in a double locked server room. According to the standards of the data protection law, all data obtained in the course of the study will be treated with discretion in order to guarantee the rights of the Participant's privacy.

Monitoring

The responsible monitor will contact and visit the clinical site regularly and will be allowed, on request, to review the various records of the study (CRFs/eCRFs and other pertinent data) provided that Participant confidentiality is maintained in accordance with local requirements and as specified in the contract. The monitor will review the study documents (e.g., CRFs) at regular intervals throughout the study, to verify the adherence to the protocol and the legibility, completeness, consistency, and accuracy of the data being entered on them. The monitor will have access to laboratory test reports and other Participant records needed to verify the entries on the CRF/eCRF. This source data verification may be carried out remotely.

Quality assurance and quality control

All Study Product used will be subjected to quality control. Quality assurance audits will be performed by the Sponsor (or any health authority) during the course of the clinical study or after its completion

Adverse Events (AE):

For purposes of this study all AEs reported will be unexpected. The causality assessment of an AE to the investigational and/or study procedure(s) product will be rated as Unrelated, Unlikely, Possible, Probable or definite using accepted criteria for clinical trials. The severity of AEs will be recorded, including the start and stop dates for each change in severity, and graded on a five-point-scale in accordance with the Common Terminology Criteria for Adverse Events. The outcome of AEs will be followed up and recorded. All Adverse Events (AEs) occurring during clinical studies will be recorded in the eCRF. During the course of the study, complete reports of all AEs will be entered in the Participants site source documents, and if applicable, on the appropriate study case report forms (CRFs). A licensed clinician will be responsible for: identifying and evaluating the severity (mild, moderate, or severe) and clinical importance of the AE, taking appropriate medical action(s), and for notifying the Sponsor immediately of an SAE as specified in the protocol and for notifying the Science Department for reporting to the IRB/IEC. For any laboratory abnormality, the PI or Sub-Investigator will make a judgement as to its clinical significance. The PI or Sub-Investigator will comply with applicable regulatory requirement(s) related to the reporting of SAEs to the IRB/IEC.

The Monitor(s) will review completed CRF data and will compare CRF entries with information recorded in the source documents. Any discrepancies or omissions in either data source will be discussed with the site personnel who should make the appropriate corrections to the documents.

ELIGIBILITY:
Inclusion Criteria:

* Be able to give written informed consent.
* Adults between 50 to 65 years inclusive.
* Has a BMI > 27 kg/m2.
* Low fibre diet, <18 g/day.
* Is in general good health, as determined by the investigator.
* Willing to consume the Study Product daily for the duration of the study.

Exclusion Criteria:

* Participants who are pregnant or wish to become pregnant during the study, or who are currently breastfeeding.
* Participants currently of childbearing potential, but not using continuous effective method of contraception.
* Metabolic disease including diabetes.
* Participants has acute or chronic gastrointestinal and/or infective disease (i.e., coeliac disease, diarrhoea, Crohn's disease, ulcerative colitis, irritable bowel syndrome, diverticulosis, stomach or duodenal ulcers, hepatitis, HIV, cancer, etc.), or with a history of such diseases.
* Have a significant acute or chronic coexisting illness such as uncontrolled hypertension, uncontrolled hyperlipidaemia, hypercoagulation, inflammatory disorders, or any condition which contraindicates, in the investigator's judgement, entry to the study.
* Smoking more than 5 cigarettes per day.
* Participant has a history of drug and/or alcohol abuse at the time of enrolment (Drinks more than nationally recommended units per week (>11 units for women; >17 units for men); alcohol/substance abuse disorder).
* Reported change in diet 30 days prior to Visit 2.
* Participants who have taken oral antibiotics 12 weeks prior to visit 2.
* Change in supplements, or major changes in lifestyle (i.e., diet, dieting, exercise level, travelling) for duration of the study.
* Has a malignant disease or any concomitant end-stage organ disease, and are severely immunocompromised (HIV positive, transplant patient, on antirejection medications, or chemotherapy or radiotherapy which, in the Investigator's judgment, contraindicates participation in the study.
* Is hypersensitive to any of the components of the Study Product.
* Has received treatment involving experimental drugs in the past 90 days and experimental supplements in the past 30 days at the discretion of the investigator.
* Any Participant who is an employee of the study site or an Atlantia Clinical Trials employee or their immediate family member or a member of their household.
* Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the study.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Effect of freeze-dried blueberry powder on the gut microbiome. | 8 weeks
  To evaluate the effect of freeze-dried blueberry powder compared to placebo, in a population comprising of overweight and obese adults on:
  - Alteration of gut microbiome function and gene count
  Change in gut microbiome function and gene count, as measured by shotgun metagenomics from baseline (Week 0) to end of intervention (Week 8).
Effect of freeze-dried blueberry powder on the gut permeability | 8 weeks
  To evaluate the effect of freeze-dried blueberry powder compared to placebo, in a population comprising of overweight and obese adults on:
  - Gut permeability
  Change in gut permeability, as measured from lactulose/mannitol ratio from baseline (Week 0) to end of intervention (Week 8).

SECONDARY OUTCOMES:
Effect of freeze-dried blueberry powder on lipid profile in a population of overweight and obese adults | 8 weeks
  evaluate the effect of freeze-dried blueberry powder compared to Placebo, in a population comprising of overweight and obese adults as assessed by:
  - Lipid profile
  Change from baseline (Week 0) to end of intervention (Week 8) on Lipid profile:
  * Total cholesterol
  * LDL
  * HDL
  * Triglycerides
Effect of freeze-dried blueberry powder on body composition in a population of overweight and obese adults | 8 weeks
  evaluate the effect of freeze-dried blueberry powder compared to Placebo on body composition in a population comprising of overweight and obese adults as assessed by:
  - Body composition
  Change from baseline (Week 0) to end of intervention (Week 8) in Body Composition measured by Bioelectrical Impedance Analysis (BIA) on:
  * Body Fat (Kg)
  * Body Fat (%)
  * Fat Mass
  * Fat Free Mass
  * Muscle Mass
Effect of freeze-dried blueberry powder on serum metabolites in a population of overweight and obese adults | 8 weeks
  evaluate the effect of freeze-dried blueberry powder compared to Placebo, in a population comprising of overweight and obese adults as assessed by:
  - Serum Metabolomics
  Serum metabolomics will be investigated by UPLC-MS using a Waters ACQUITY ultra-performance liquid chromatography (UPLC) and a Thermo Scientific Q-Exactive high resolution/accurate mass spectrometer interfaced with a heated electrospray ionization (HESI-II) source and Orbitrap mass analyzer operated at 35,000 mass resolution. Metabolites will be annotated by the UPLC-MS operator, providing a list of chemical compounds and their concentrations.
Effect of freeze-dried blueberry powder on urine and faecal metabolites in a population of overweight and obese adults | 8 weeks
  evaluate the effect of freeze-dried blueberry powder compared to Placebo, in a population comprising of overweight and obese adults as assessed by:
  Change from baseline (Week 0) to end of intervention (Week 8) on:
  * Urine metabolic markers
  * Faecal metabolic markers
  Urine and Faecal metalbolites will be measured as for serum metabolites (UPLC-MS)
Effect of freeze-dried blueberry powder on faecal bile acid metabolites in a population of overweight and obese adults | 8 weeks
  evaluate the effect of freeze-dried blueberry powder compared to Placebo, in a population comprising of overweight and obese adults as assessed by:
  Change from baseline (Week 0) to end of intervention (Week 8) on:
  - Faecal bile acid metabolites
  Faecal levels of bile acids will be measured by targeted metabolomics
Effect of freeze-dried blueberry powder on polyphenol metabolites in a population of overweight and obese adults | 8 weeks
  evaluate the effect of freeze-dried blueberry powder compared to Placebo, in a population comprising of overweight and obese adults as assessed by:
  Change from baseline (Week 0) to end of intervention (Week 8) on:
  - Polyphenol metabolites
  Polyphenol metabolites will be identified by HPLC or UPLC-MS based on reference to standard compounds or mass/charge reference libraries.

CONTACTS AND LOCATIONS:
Overall Officials: Paul W. O'Toole, Prof., Study Director — University College Cork; Timothy Dinan, Prof., Principal Investigator — Atlantia Clinical Trials
Locations (1):
- Atlantia Food Clinical Trials, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No